CLINICAL TRIAL: NCT03323398
Title: A Phase 1/2, Open-Label, Multicenter, Dose Escalation and Efficacy Study of mRNA-2416, a Lipid Nanoparticle Encapsulated mRNA Encoding Human OX40L, for Intratumoral Injection Alone or in Combination With Durvalumab for Patients With Advanced Malignancies
Brief Title: Dose Escalation and Efficacy Study of mRNA-2416 for Intratumoral Injection Alone and in Combination With Durvalumab for Participants With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was halted prematurely because the efficacy endpoints were not met for either treatment arm.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-2416-P101
Record Dates: First submitted 2017-10-23; First posted 2017-10-27 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-06

CONDITIONS: Relapsed/Refractory Solid Tumor Malignancies or Lymphoma; Ovarian Cancer
Keywords: mRNA-2416; OX40 ligand; OX40L; Moderna
MeSH Terms: conditions — Recurrence; Lymphoma; Ovarian Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: mRNA-2416 Alone (Experimental): Participants will be administered mRNA-2416 through an intratumoral injection at the applicable dose on Days 1 and 15 for six 28-day cycles.
  Interventions: Biological: mRNA-2416
- Arm B: mRNA-2416 in Combination with Durvalumab (Experimental): Participants will be administered mRNA-2416 through an intratumoral injection at the applicable dose on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 6 in combination with durvalumab through an intravenous infusion at a fixed dose on Day 1 of Cycles 1 through 6. The duration for each cycle is 28 days.
  Interventions: Biological: mRNA-2416; Biological: Durvalumab

INTERVENTIONS:
Biological: mRNA-2416 — mRNA encoding human OX40L
Biological: Durvalumab — PD-L1 inhibitor
  Arms: Arm B: mRNA-2416 in Combination with Durvalumab

SUMMARY:
This clinical study will assess the safety and tolerability of escalating doses of mRNA-2416 alone and in combination with administered fixed doses of durvalumab in participants with relapsed/refractory solid tumor malignancies or lymphoma, as well as the objective response rate (ORR) of mRNA-2416 alone or in combination with durvalumab in ovarian cancer based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The applicable dose of mRNA-2416 will be injected directly into the participant's tumor (intratumoral) and the applicable dose of durvalumab will be administered intravenously.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/2, open-label, multicenter, dose escalation and efficacy study designed to determine the safety and tolerability of repeated intratumoral injections of mRNA-2416 alone (Arm A) and in combination with intravenously administered durvalumab (Arm B) in participants with advanced relapsed/refractory solid tumor malignancies or lymphoma and to assess the ORR of mRNA-2416 alone and in combination with durvalumab in ovarian cancer based on RECIST v1.1. The study includes 2 treatment arms (mRNA-2416 monotherapy [Arm A],and mRNA-2416 + durvalumab [Arm B]), each arm of the study consists of a Dose Escalation period in non-visceral lesions followed by a Dose Confirmation period in visceral lesions and an Expansion period (Arm B only) in participants with ovarian cancer at the MTD/RDE as determined by the Dose Escalation period. Once the expected maximum tolerated dose/recommended dose for expansion (MTD/RDE) has been cleared in Dose Escalation for Arm A, Dose Escalation for Arm B will begin with mRNA-2416 at 1 dose level lower than the Arm A MTD/RDE.

Following completion of 6 cycles of mRNA-2416 + durvalumab (Arm B), participants may continue with durvalumab alone until disease progression, unacceptable toxicity, or 24 months of treatment (total), whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to completing any study-specific procedure
* Dose Escalation and Dose Confirmation Periods: Histologically- or cytologically-confirmed advanced/metastatic solid tumor or lymphoma by pathology report and who has received, or been intolerant to, all approved therapies
* Dose Expansion Period: Histologically or cytologically confirmed diagnosis of: epithelial cancer of the ovary, fallopian tube, or peritoneum which is platinum resistant or platinum refractory. Participants must have received at least 2 prior lines of therapy. Participants with known Breast Cancer gene 1 (BRCA) mutation positive must have been treated with and progressed on at least 1 prior poly[ADP-ribose] polymerase inhibitor (PARPi)
* Lesions for intratumoral injection and biopsies:

  * Dose Escalation: A minimum of one lesion that is easily accessible for injection where easily accessible is defined as a cutaneous or subcutaneous mass that is palpable and/or visualizable by ultrasound
  * Dose Confirmation: A minimum of one visceral lesion injectable with ultrasound or computer tomography (CT) guidance and that is not encasing or abutting major vascular structures or are in a location that are considered high risk for AEs by the enrolling physician
  * Dose Expansion: A minimum of one lesion amenable to injection (either non-visceral or visceral). Participants must have a tumor lesion amenable to biopsy and consent to a pre-treatment and an on-treatment biopsy. For participants with only one lesion amenable to injection, biopsy, and RECIST assessment, the lesion must be ≥2 centimeters (cm)
  * Biopsy Cohort Enrichment: Participants must have a tumor lesion amenable to biopsy and consent to a pre-treatment and an on-treatment biopsy
* All lesion(s) targeted for the initial injection must be ≥0.5 cm on longest diameter, be at least 5 mm thick, and have distinct borders based on exam or imaging, not close to critical structures such as major vessels, nerves, or airways
* Participants must have measurable disease as determined by RECIST v1.1 (solid tumors) or Cheson 2014 criteria (lymphomas).

  - Dose Expansion: Participants must have at least 1 measurable lesion per RECIST v1.1 which has not been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate hematological and biological function
* Adequate thyroid function: Thyroid-stimulating hormone within normal range.
* Female participants of childbearing potential must have a negative serum pregnancy test during screening.
* Male and female participants must agree to use a highly reliable method of birth control.
* Must have life expectancy of at least 12 weeks
* Body weight >30 kilograms (kg)

Exclusion Criteria:

* Active central nervous system tumors or metastases
* Treatment with chemotherapy, radiation (local radiation for palliative care is permitted), hormonal anti-cancer treatment, or biologic therapy <14 days prior to the first day of study treatment (Cycle 1 Day 1 [C1D1]). Treatment with any other investigational agent or treatment with any anti-cancer monoclonal antibody, immunostimulant, or vaccine <28 days prior to C1D1
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Participants with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
  * Participants with irreversible toxicity not reasonably expected to be exacerbated by the treatment with durvalumab may be included only after consultation with the Study Physician
* Has active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [for example, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [for example, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis]). The following are exceptions to this criterion:

  * Participants with vitiligo or alopecia
  * Participants with hypothyroidism (for example, following Hashimoto syndrome) stable on hormone replacement
  * Participants with any chronic skin condition that does not require systemic therapy
  * Participants without active disease in the last 5 years may be included but only after consultation with the Moderna medical monitor
  * Participants with celiac disease controlled by diet alone
* Has a history of primary immunodeficiency, allogenic solid organ transplantation, or tuberculosis
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Participants, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment.
* History of human immunodeficiency virus infection
* Active/chronic hepatitis B or C
* Any of the following cardiac abnormalities:

  * Medically uncontrolled hypertension
  * New York Heart Association Class III or IV cardiac disease
  * Myocardial infarction within prior 6 months
  * Unstable angina
  * Unstable arrhythmias or mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 milliseconds (ms) calculated from 3 electrocardiograms (ECGs) (within 15 minutes at 5 minutes apart)
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Females who are pregnant or breastfeeding
* Any other unstable or clinically significant concurrent medical condition (for example, substance abuse, psychiatric illness/social situations, uncontrolled intercurrent illness including active infection, arterial thrombosis, symptomatic pulmonary embolism, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea) that would, in the opinion of the investigator, jeopardize the safety of a participant, impact their expected survival through the end of the study participation, and/or impact their ability to give written informed consent or comply with the protocol
* For participants who have received prior anti-programmed death 1 (PD-1) or anti-programmed death ligand 1 (PD-L1) therapy, a participant must not have experienced any of the following:

  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
* Must not have experienced a Grade ≥3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. Note: Participants with endocrine AEs of Grade ≤2 are permitted to enroll if they are stable while maintained on appropriate replacement therapy and are asymptomatic.
* Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of >10 milligrams (mg) prednisone or equivalent per day.
* Has an active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a history of leptomeningeal carcinomatosis.
* Has involvement in the planning and/or conduct of the study.
* Must not plan to donate blood or blood components while participating in this study and through 90 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Northwestern Memorial Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Women & Infants Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to include participants with lymphoma in the study, but none of the enrolled participants had lymphoma.
Pre-assignment Details: 79 participants were enrolled into the study. 18 participants screen failed, and so 61 participants were randomized. Data are presented for the 61 randomized participants.
Groups:
- Arm A, Dose Escalation: mRNA-2416 1.0 Milligrams (mg) Alone: Participants were administered mRNA-2416 through an intratumoral injection at a dose of 1.0 mg on Days 1 and 15 for six 28-day cycles.
- Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone: Participants were administered mRNA-2416 through an intratumoral injection at a dose of 2.0 mg on Days 1 and 15 for six 28-day cycles.
- Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone: Participants were administered mRNA-2416 through an intratumoral injection at a dose of 4.0 mg on Days 1 and 15 for six 28-day cycles.
- Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone; Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone: Participants were administered mRNA-2416 through an intratumoral injection at a dose of 8.0 mg on Days 1 and 15 for six 28-day cycles.
- Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab: Participants were administered mRNA-2416 through an intratumoral injection at 4.0 mg on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 6 and durvalumab through an intravenous infusion at a fixed dose (1500 mg, except for participants whose weight fell to ≤30 kilograms [kg] received a weight-based dose at 20 mg/kg) on Day 1 of Cycles 1 through 6. The duration of each cycle was 28 days.
- Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab; Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab: Participants were administered mRNA-2416 through an intratumoral injection at 4.0 mg on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 6 and durvalumab through an intravenous infusion at a fixed dose (1500 mg, except for participants whose weight fell to ≤30 kg received a weight-based dose at 20 mg/kg) on Day 1 of Cycles 1 through 6. The duration of each cycle was 28 days.
- Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab: Participants were administered mRNA-2416 through an intratumoral injection at 2.0 mg on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 6 and durvalumab through an intravenous infusion at a fixed dose (1500 mg, except for participants whose weight fell to ≤30 kg received a weight-based dose at 20 mg/kg) on Day 1 of Cycles 1 through 6. The duration of each cycle was 28 days.
Period: Overall Study
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 Milligrams (mg) Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab
Started | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
Received At Least 1 Dose of Study Drug | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
Completed | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 7
Not Completed | 9 | 11 | 10 | 2 | 1 | 3 | 2 | 1 | 8
Not completed — Other than Specified | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 6 | 2 | 2 | 1 | 2 | 0 | 0 | 6
Not completed — Received Alternative Anticancer Therapy | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant was Put on Hospice | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Discontinued Following Discussion with Physician | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all enrolled participants who received any amount of study drug. Participants were included in the dose cohort corresponding to the dose level they actually received. No baseline characteristics data is reported for Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone or Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab to maintain participant confidentiality.
Groups:
- Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone: Participants were administered mRNA-2416 through an intratumoral injection at a dose of 1.0 mg on Days 1 and 15 for six 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab | Total
Number analyzed (Participants) | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No baseline characteristics data is reported for Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone or Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab to maintain participant confidentiality.
  years
    number analyzed (Participants) | 11 | 12 | 12 | 3 | 0 | 3 | 3 | 0 | 15 | 59
    (all) | 64.6 (7.55) | 59.8 (17.40) | 64.4 (11.18) | 69.3 (5.69) |  | 66.0 (7.81) | 50.3 (23.59) |  | 64.1 (64.0) | 63.1 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No baseline characteristics data is reported for Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone or Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab to maintain participant confidentiality.
  Participants
    number analyzed (Participants) | 11 | 12 | 12 | 3 | 0 | 3 | 3 | 0 | 15 | 59
    Female | 4 | 4 | 8 | 1 |  | 0 | 2 |  | 15 | 34
    Male | 7 | 8 | 4 | 2 |  | 3 | 1 |  | 0 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: No baseline characteristics data is reported for Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone or Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab to maintain participant confidentiality.
  Participants
    number analyzed (Participants) | 11 | 12 | 12 | 3 | 0 | 3 | 3 | 0 | 15 | 59
    Hispanic or Latino | 0 | 1 | 3 | 0 |  | 0 | 0 |  | 0 | 4
    Not Hispanic or Latino | 11 | 11 | 9 | 3 |  | 3 | 3 |  | 15 | 55
    Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: No baseline characteristics data is reported for Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone or Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab to maintain participant confidentiality.
  Participants
    Race: number analyzed (Participants) | 11 | 12 | 12 | 3 | 0 | 3 | 3 | 0 | 15 | 59
    Race: White | 10 | 11 | 10 | 3 |  | 3 | 2 |  | 14 | 53
    Race: Other | 0 | 1 | 0 | 0 |  | 0 | 0 |  | 0 | 1
    Race: Not Reported | 1 | 0 | 2 | 0 |  | 0 | 0 |  | 1 | 4
    Race: Black or African American | 0 | 0 | 0 | 0 |  | 0 | 1 |  | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs: assessed by Investigator as unrelated to disease, disease progression, intercurrent illness, or concomitant medications; at least possibly related to study drug; and occurred within first 28 days of the study. DLTs in Arm A participants: Grade (Gr)3 adverse events (AEs) (except Gr3 thrombocytopenia lasting <7 days/Gr3 neutropenia without fever or lasting <7 days) and any Gr4/5 toxicity. DLTs (criteria assessed by Investigator) participants in Arm B: diarrhea/colitis; pneumonitis; hepatitis; rash; peripheral neuromotor syndromes; myocarditis; myositis/polymyositis; endocrinopathies involving thyroid, pituitary glands, or adrenal insufficiency; type I diabetes mellitus; nephritis; elevated amylase/lipase pancreatitis; all other immunemediated/nonimmunemediated AEs; infusion-related reactions; any Gr≥3 immune/nonimmune AE except vitiligo/alopecia; neutropenia Gr≥3 with fever/Gr4 lasting >7 days; Gr≥3 thrombocytopenia and significant bleeding; Gr4 thrombocytopenia; and Gr4 anemia.
Time Frame: Days 1-28 (Cycle 1)
Population: The Safety Set included all enrolled participants who received any amount of study drug. Participants were included in the dose cohort corresponding to the dose level they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit: Participants were administered mRNA-2416 through an intratumoral injection at 4.0 mg on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 through 6 and durvalumab through an intravenous infusion at a fixed dose (1500 mg, except for participants whose weight fell to ≤30 kilograms [kg] received a weight-based dose at 20 mg/kg) on Day 1 of Cycles 1 through 6. The duration of each cycle was 28 days.
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With a Treatment-Emergent AEs (TEAE) or a Serious AE
Description: An AE is any adverse experience in a participant administered a study drug, whether or not it is considered drug related, that occurred during study participation. This would include any side effect, injury, toxicity, sensitivity reaction, intercurrent illness, or sudden death. Conditions that started before study entry were reported as an AE if the frequency, intensity, or character of the condition worsened during the study. A TEAE was defined as any AE that newly appeared, increased in frequency, or worsened in severity following initiation of study drug. A serious AE (SAE) was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 up to 90 days after the last dose of study treatment (maximum exposure=26.3 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
Participants
  TEAE | 10 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
  SAE | 3 | 6 | 7 | 2 | 1 | 2 | 2 | 1 | 11

3. Primary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as the percentage of participants in the Activity Evaluable Set with best overall response of Partial Response (PR) or better, where the denominator was the number of participants with solid tumor. Solid tumor response was assessed by Investigators based on RECIST version 1.1 (complete response [CR], PR, stable disease [SD], progressive disease [PD], or not evaluable), and based on Immune-related Response Criteria (irRC) (immune-related CR, immune-related PR, immune-related SD, immune-related PD, or not evaluable). The 95% confidence interval (CI) was based on the Clopper-Pearson exact test.
Time Frame: Day 1 through 6 months after the last dose of study treatment, or until disease progression, whichever occurred first (maximum exposure=26.3 weeks)
Population: The Activity Evaluable Set included all enrolled participants who received any amount of study drug and had at least 1 tumor response evaluation. Participants were included in the dose cohort to which they were enrolled. One of the participants excluded from this analysis for the arm labeled "Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab" was excluded due to a diagnosis of cervical cancer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 8 | 9 | 8 | 3 | 1 | 2 | 3 | 1 | 13
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5] | 7.7 [0.2 to 36.0]

4. Secondary Outcome: Duration of Response in Participants With Ovarian Cancer (RECIST Version 1.1)
Description: Duration of response was defined as the time from first response (PR or better, as assessed by Investigators based on RECIST version 1.1) to first occurrence of a disease progression. Participants who never achieved a response were excluded from this analysis. DOR (days) = date of event/censoring - date of first response + 1. Duration of response could only be calculated if more than 1 participant had a PR. Since only 1 participant had a PR, the duration of response could not be calculated.
Time Frame: Day 1 through 6 months after last dose of study treatment, or until disease progression, whichever occurred first (maximum exposure=26.3 weeks)
Population: The Activity Evaluable Set included all enrolled participants who received any amount of study drug and had at least 1 tumor response evaluation. Participants were included in the dose cohort to which they were enrolled. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure. Since only 1 participant had a PR, the duration of response could not be calculated.
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Disease Control Rate in Participants With Ovarian Cancer (RECIST Version 1.1)
Description: Disease control rate (DCR) was defined as the percentage of participants in the Activity Evaluable Set with best overall response of PR or better, or SD ≥55 days (from the first dose date to the last SD assessment, and without PD between), where the denominator is the number of participants with solid tumor. Solid tumor response was assessed by investigators based on RECIST version 1.1 (CR, PR, SD, PD, or not evaluable), and based on irRC (immune-related CR, immune-related PR, immune-related SD, immune-related PD, or not evaluable). The 95% CI was based on the Clopper-Pearson exact test.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 8 | 9 | 8 | 3 | 1 | 2 | 3 | 1 | 13
percentage of participants | 50.0 [15.7 to 84.3] | 33.3 [7.5 to 70.1] | 12.5 [0.3 to 52.7] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 100.0 [2.5 to 100.0] | 15.4 [1.9 to 45.4]

6. Secondary Outcome: Number of Participants With Anti-OX40L Antibodies
Description: Data are presented for number of participants with anti-OX40L antibodies. OX40L is the protein translated by the drug product.
Time Frame: Cycle (C) 1 Day (D) 1, C1D15, C2D1, C3D1, C3D15, C4D1, C5D1, C6D1, C6D15, End of Treatment (maximum exposure=26.3 weeks); Cycle =28 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and DurvalumabEdit
Number analyzed (Participants) | 11 | 12 | 12 | 3 | 1 | 3 | 3 | 1 | 15
Participants
  C1D1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  C3D1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  C3D15 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  C4D1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  C5D1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  C6D1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C6D15 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  End of Treatment | 4 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 90 days after the last dose of study treatment (maximum exposure=26.3 weeks)
Description: The Safety Set included all enrolled participants who received any amount of study drug. Participants were included in the dose cohort corresponding to the dose level they actually received. The data reported for "All-Cause Mortality" included the participants who were discontinued due to "Death" and the participant who was discontinued due to "Intent to go to a Hospice" who subsequently died.
Arm/Group | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab | Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab
All-Cause Mortality (participants affected / at risk) | 4/11 | 6/12 | 3/12 | 2/3 | 1/1 | 2/3 | 0/3 | 0/1 | 6/15
Serious Adverse Events (participants affected / at risk) | 3/11 | 6/12 | 7/12 | 2/3 | 1/1 | 2/3 | 2/3 | 1/1 | 11/15
Other Adverse Events (participants affected / at risk) | 10/11 | 12/12 | 12/12 | 3/3 | 0/1 | 3/3 | 3/3 | 1/1 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone (N=11) | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone (N=12) | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone (N=12) | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone (N=3) | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone (N=1) | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab (N=3) | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab (N=3) | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab (N=1) | Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab (N=15)
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Dose Escalation: mRNA-2416 1.0 mg Alone (N=11) | Arm A, Dose Escalation: mRNA-2416 2.0 mg Alone (N=12) | Arm A, Dose Escalation: mRNA-2416 4.0 mg Alone (N=12) | Arm A, Dose Escalation: mRNA-2416 8.0 mg Alone (N=3) | Arm A, Dose Confirmation: mRNA-2416 8.0 mg Alone (N=1) | Arm B, Dose Escalation: mRNA-2416 4.0 mg and Durvalumab (N=3) | Arm B, Dose Confirmation: mRNA-2416 4.0 mg and Durvalumab (N=3) | Arm B, Dose Expansion: mRNA-2416 2.0 mg and Durvalumab (N=1) | Arm B, Dose Expansion: mRNA-2416 4.0 mg and Durvalumab (N=15)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 6
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 4
Flushing (Vascular disorders) | 2 | 3 | 4 | 1 | 0 | 0 | 2 | 0 | 3
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Essential hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 4 | 0 | 0 | 1 | 2 | 1 | 11
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 7
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 0 | 0 | 0 | 1 | 0 | 7
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue pigmentation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 3 | 6 | 1 | 0 | 0 | 2 | 1 | 12
Pyrexia (General disorders) | 3 | 3 | 3 | 1 | 0 | 0 | 2 | 1 | 8
Injection site pain (General disorders) | 1 | 5 | 5 | 0 | 0 | 1 | 0 | 1 | 8
Oedema peripheral (General disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 4
Influenza like illness (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Injection site erythema (General disorders) | 0 | 4 | 2 | 2 | 0 | 1 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 5
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 5
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Action tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial spasm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bladder irritation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site vesicles (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Antiphospholipid antibodies positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nerve root injury sacral (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was halted prematurely because the efficacy endpoints were not met for either treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03323398/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT03323398/SAP_001.pdf